CLINICAL TRIAL: NCT06798051
Title: A Single-dose, Fasting, Randomized, Open-label, Two-treatment, Three-period, Partially-replicated, Reference-corrected Crossover Bioequivalence Study of Roxithromycin Tablets in Healthy Subjects
Brief Title: Bioequivalence Study of Two Roxithromycin Tablets in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The Affiliated Hospital Of Guizhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: KL288-1-BE-01
Record Dates: First submitted 2025-01-14; First posted 2025-01-29 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Bioequivalence of Roxithromycin Tablets From Two Different Manufacturers
MeSH Terms: interventions — Roxithromycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- A group T-R-R (Experimental)
  Interventions: Drug: Roxithromycin tablets 150mg
- B group R-T-R (Experimental)
  Interventions: Drug: Roxithromycin tablets 150mg
- C group R-R-T (Experimental)
  Interventions: Drug: Roxithromycin tablets 150mg

INTERVENTIONS:
Drug: Roxithromycin tablets 150mg — Oral roxithromycin tablets，150mg Once every seven days，One cycle T drug, two cycles R drug

SUMMARY:
Roxithromycin is used for the treatment of pharyngitis and tonsillitis caused by Streptococcus pyogenes, sinusitis, otitis media, acute bronchitis, acute exacerbations of chronic bronchitis, and pneumonia caused by Mycoplasma pneumoniae or Chlamydia pneumoniae; urethritis and cervicitis caused by Chlamydia trachomatis; and skin and soft tissue infections caused by susceptible bacteria.

The purpose of this study was to evaluate the bioequivalence of roxithromycin tablets from two different manufacturers after fasting administration in healthy subjects and to observe the safety of the test and reference preparations in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Chinese healthy adults over 18 years old ( including 18 years old ) ;
* Weight : male ≥ 50.0kg, female ≥ 45.0kg and body mass index ( BMI ) :

19.0 ~ 26.0kg / m2 ( including boundary value, BMI = weight ( kg ) / height ( m ) 2 ) ;

* Understand and sign the informed consent, volunteer to participate in this study ;
* Be able to communicate well with the researchers and complete the study in accordance with the provisions of the study.

Exclusion Criteria:

* There is a history of diseases such as cardiovascular system, respiratory system, digestive system, endocrine system, nervous / mental system, blood and lymphatic system, skeletal muscle system, family genetic disease history and so on;
* Patients who had undergone major surgery within 1 year before screening and were judged not suitable for enrollment by the researchers;
* Comprehensive physical examination, vital signs, 12-lead electrocardiogram, laboratory tests [ including blood routine, urine routine, blood biochemistry, coagulation function, blood pregnancy ( only female subjects ) ], etc., suggested that there were abnormalities judged by the researchers as clinically significant ;
* electrolyte potassium < 3.5mmol / L or magnesium < 0.75mmol / L in blood biochemistry ;
* hepatitis B surface antigen ( HBsAg ), hepatitis B e antigen ( HBeAg ), hepatitis C antibody ( HCV-Ab ), human immunodeficiency virus antibody ( HIV-Ab ), treponema pallidum antibody ( TP-Ab ) any test results positive ;
* the existence of researchers judged to have clinical significance of food, drug allergy or other allergic disease history ( asthma, urticaria, eczematous dermatitis, etc. ) or the product and its excipients or its analogues allergy ;
* Patients who used any drugs that interact with roxithromycin within 30 days before screening ( such as contraceptives, ergotamine/dihydroergotamine, theophylline, anticoagulants, digoxin and other cardiac glycosides, midazolam, cyclosporine, drugs that can prolong QT interval [antidepressants ( such as citalopram ), antiarrhythmic drugs ( such as sotalol, amiodarone ), cisapride, antipsychotics ( such as clozapine

  * antibiotics ( such as erythromycin ) ] ;
* who had used any drug within 2 weeks before screening, and was judged by the researcher to be likely to affect the evaluation results of this study ;
* Patients with a history of drug abuse / drug dependence or positive urine screening within 12 months before screening ;
* Patients who drank more than 14g alcohol per week ( 1 unit = 360ml beer or 45ml alcohol with 40 % alcohol or 150ml wine ) within 6 months before screening, or who could not give up drinking during the trial, or who were positive for alcohol breath test ;
* patients who had long-term excessive drinking ( more than 8 cups a day, 1 cup = 250ml ) of tea, coffee or caffeine-containing beverages ;
* Smoking ≥ 3 cigarettes per day within 3 months before screening or those who could not guarantee to give up smoking during the trial ;
* Patients who participated in other drug clinical trials and took research drugs within 3 months before screening ( the last visit time of the last trial was calculated as the start time ) ;
* Screening for blood donation or blood products or massive bleeding > 200ml or 1 unit within the first 3 months, or planning to donate blood or blood components during the study period ;
* Do not agree to avoid the use of tobacco ( including any nicotine-containing smoking cessation products such as nicotine lozenges, nicotine gum ), wine or xanthine, grapefruit, caffeine ( such as coffee, strong tea, chocolate, etc. ) drinks or food ( such as animal liver, mango, pitaya, etc. ), or to avoid strenuous exercise, or to avoid other factors affecting drug absorption, distribution, metabolism, excretion, etc. ;
* Pregnant or lactating women, or those with positive pregnancy test results before the test ; male subjects or female subjects were unwilling to take one or more non-drug contraceptive measures ( such as complete abstinence, contraceptive ring, partner ligation, etc. ) during the trial, or had sperm / egg donation plans or male subjects ( or their partners ), female subjects had fertility plans ( from the signing of informed consent to 3 months after the last administration ) ;
* patients with difficulty in venous blood collection or fainting ;
* tablet swallowing difficulties ;
* those who have special requirements for diet, cannot abide by the diet provided and the corresponding regulations ;
* Subjects who were considered inappropriate to participate in this clinical study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2019-06-03 (Actual); Primary Completion 2019-08-06 (Actual); Study Completion 2019-09-03 (Actual)

PRIMARY OUTCOMES:
maximum observed serum or plasma concentration | 3 day
  The with-subject standard deviation of the pharmacokinetic parameter Cmax of the reference preparation was calculated and the bioequivalence was analyzed according to the bioequivalence evaluation criteria.
area under the serum or plasma concentration-time curve from 0 to t | 3 day
  The with-subject standard deviation of the pharmacokinetic parameter AUC0-t of the reference preparation was calculated and the bioequivalence was analyzed according to the bioequivalence evaluation criteria.
area under the serum or plasma concentration-time curve from 0 to infinity | 3 day
  The with-subject standard deviation of the pharmacokinetic parameter AUC0- ∞ of the reference preparation was calculated and the bioequivalence was analyzed according to the bioequivalence evaluation criteria.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Trials Center, The Affiliated Hospital of Guizhou Medical University, Guiyang, China